CLINICAL TRIAL: NCT04019639
Title: Clinical Trial for the Efficacy and Safety of Paste Type Acellular Dermal Matrix in Chronic Wound Healing
Brief Title: Efficacy of Paste Type Acellular Dermal Matrix(CG Paste) in Chronic Wound Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government); Hanyang University (Other); St Vincent's Hospital (Other)
Responsible Party: Principal Investigator, Sang Wha Kim, assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-02
Record Dates: First submitted 2019-06-03; First posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Chronic Wound
Keywords: ADM; acellular dermal matrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CG Paste+EasyFoam (Experimental): The subjects assigned to the test group through random assignment will receive the wound treatment by applying CG Paste and EasyFoam. CG Paste is a medical device currently marketed in CGBio.It is a free-flowing, acellular allogeneic dermis processed from human tissue skin, and then granulated and homogenized. This increases the water content and viscosity of the micronized ADM particles mixed with the gelatin sol carrier to protect the wound area and maintain the wet environment by applying to the desired wound area.It contains collagen, elastin and various growth factors in the dermis and has excellent tissue compatibility compared to the heterogeneous or synthetic material, so that the immune rejection is hardly observed in the graft site.
  It also contains collagen, elastin, fibronectin, laminin, and proteoglycans, which are components of the human skin, to help the interaction between normal cells and extracellular matrix.
  Interventions: Device: application of CG Paste+EasyFoam
- EasyFoam (Active Comparator): Subjects randomly assigned to the control group receive EasyFoam treatment for wound healing.
  The foam has excellent moisture permeability, absorbs a large amount of exudates, and prevents scar formation to minimize scar formation.
  Interventions: Device: application of EasyFoam

INTERVENTIONS:
Device: application of CG Paste+EasyFoam — Prior to application of CG paste, sharp debridement can be performed first in the operating room under local anesthesia or general anesthesia. After this, hemostasis is performed by an electrocoagulator and the medical device is applied to the affected area. During the procedure, remove the packaging material and remove the syringe to remove the protective cap in front of the syringe. Slowly push the syringe plunger and apply the contents to the area where you want to use. Depending on the location and size of the wound area, an injection cap can be used. Apply CG paste and apply Easyfoam to finish the dressing.
  Arms: CG Paste+EasyFoam
Device: application of EasyFoam — Prior to applying EasyFoam, sharp debridement can be performed first in the operating room under local anesthesia or general anesthesia. Marginal resection is performed until the necrotic tissue is removed sufficiently and pin point bleeding is seen on the wound. After that, hemostasis is done with an electrocoagulator and EasyFoam is applied to the affected area.
  Arms: EasyFoam

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of wound sizing and completeness in chronic window treatment, and to confirm the superiority of area reduction in CG Paste and form-dressing as compared to form-dressing alone groups and CG Paste and form-dressing companion groups.

DETAILED DESCRIPTION:
wound refers to a condition in which the skin is damaged by a cause. In general, open wound rather than closed wound requires active treatment. It is important to make sure that the wound are cured early and through proper treatment. If the wound is open for a long time, secondary complications such as infection can occur and are easy to transition to chronic wound. Chronic wound refers to an idea that does not heal after a period of time after a normal wound healing process, which is usually defined as if it does not heal for more than three to four weeks. 1. These chronic wound include diabetic foot ulcer, pressure ulcer, vascular ulcer, etc. In addition, with the recent aging of the population, the proportion of elderly patients increases, and the proportion of chronic wound where even simple surgical wound does not heal normally, resulting in increased expenditure on health care and decreased quality of life for patients.

Biotechnical dermal transplantation material, including acellular dermal matrix, are known to be more effective in wound healing than conventional wound treatments.

The mechanism of action of acellular matrices including acellular dermal matrix, is as follows: 1) it functions as a support for cell growth and granulation tissue formation, 2) has receptors capable of attaching to fibroblasts, 3) induction of angiogenesis, 4) chemoattractant activity of vascular endothelial cells, 5) role of providing various growth factors, and temporary storage function.

Unlike other products generally known as CG paste, the acellular allo-dermal matrix product to be used in this study is made into a paste type for ease of use after freeze-drying and granulation process after undergoing the process of degreasing of the same kind of dermis . Conventional sheet-type products can not be applied to curved wounds, they must be cut and rehydrated during use, while CG paste is easy to apply to curved wounds and can be applied directly to the desired wound area without rehydration It is expected to be a ready-to-use product with similar clinical effects to existing acellular allo-dermal matrix.

The purpose of this study is to evaluate the efficacy and safety of wound sizing and completeness in chronic window treatment, and to confirm the superiority of area reduction in CG Paste and form-dressing as compared to form-dressing alone groups and CG Paste and form-dressing companion groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 19 years
* Patients with skin defect from full-thickness skin defect to bone exposure level after debridement of wound
* Chronic wounds that have not been healed despite adequate treatment for more than 3 weeks after wounding
* At the time of the study, patients with a wound size of 4 cm 2 or more

Exclusion Criteria:

* Patients with superficial or partial thickness skin defect
* osteomyelitis patient
* An undermining wound, tunneling wound, which can not measure the exact depth, can be used if the wound is open wound due to debridement of wound.
* Patients who exceeded 12% of HbA1c within 3 months before participating in the study
* Patients with serum creatinine concentration of 3.0 mg / dL or more within 30 days before the study
* Patients who have applied other medical devices and growth factors for wound healing within 30 days before participating in the study
* Patients with lesion infections (available after infection treatment)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-04-05 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
wound reduction rate | 12 weeks
  At 12 weeks after the application of the medical device, the wound reduction At 12 weeks after the application of the medical device, the wound reduction rate

SECONDARY OUTCOMES:
Complete healing rate | 12 weeks
  Complete healing rate after 12 weeks of medical device application
  * Definition of complete healing: A complete healing is defined as a state in which the skin is completely reepithelialized and the skin is completely closed. Additional operations such as skin grafting, flap surgery, primary suture, etc. are not performed.
  (definition of complete healing:
Period of time to complete healing | The period to complete healing(through study completion, an average of 12 weeks)
  Period of time from medical device application to complete healing
  * Definition of complete healing: A complete healing is defined as a state in which the skin is completely reepithelialized and the skin is completely closed. Additional operations such as skin grafting, flap surgery, primary suture, etc. are not performed.
Step of granulation tissue | 12 weeks
  Step for 12weeks of granulation tissue (The steps of granulation tissues are visualized by the following criteria, and the steps are recorded separately from A-E)
  * A: Skin intact or partial thickness wound
  * B: Bright, beefy red; 75% to 100% of wound filled & or tissue overgrowth
  * C: right, beefy red; < 75% & > 25% of wound filled
  * D: Pink, &/or dull, dusky red & or fills ≤ 25% of wound
  * E: No granulation tissue present
The time it took to reach granulation tissue formation | The period of time required for granulation tissue formation to reach 100% (through study completion, an average of 12 weeks)
  The period of time required for granulation tissue formation to reach 100%
Level of tissue exposed after 12 weeks of medical device application | 12 weeks
  After 12 weeks of medical device application, the level of exposed tissue is divided into partial thickness skin, full thickness skin, subcutaneous, deep fascia, muscle, tendon, bone, and joint, and the distribution is compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Wha Kim, Ph.D, Principal Investigator — Seoul National University Hospital; Youn Hwan Kim, Ph.D, Principal Investigator — Hanyang University; Hyung Sup Shim, Ph.D, Principal Investigator — St Vincent's Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea